CLINICAL TRIAL: NCT03806348
Title: Early Resuturing Versus Expectant Management Following Perineal Wound Dehiscence: a Randomised Controlled Trial
Brief Title: Early Resuturing Versus Expectant Management Following Perineal Wound Dehiscence Among Women Who Had a Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Marion Ek, Senior Consultant, Stockholm South General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Paris2018
Record Dates: First submitted 2018-11-29; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Wound; Perineal Rupture, Dehiscence
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resuturing (Experimental): Early resuturing of perineal wound dehiscence. Antibiotics: Amoxicillin 500 mg, Clavulanic Acid 125 mg and Metronidazole 400 mg by mouth, every 8 hours, for at least 6 Days.
  Interventions: Procedure: Resuturing
- Conservative treatment (No Intervention): Antibiotics: Amoxicillin 500 mg, Clavulanic Acid 125 mg and Metronidazole 400 mg by mouth, every 8 hours, for at least 6 Days.

INTERVENTIONS:
Procedure: Resuturing — Early reconstruction of the perineal body after wound dehiscence within two weeks of delivery.
  Arms: Resuturing

SUMMARY:
Women who deliver their baby vaginally often suffer from a perineal wound. The wound is after being sutured sometimes dehisced after days up to a few weeks and this study will investigate whether it is better to resuture early or leave the rupture for secondary healing.

DETAILED DESCRIPTION:
140 women will be included in the trial, 70 women will be randomized to resuturing and 70 women will be randomized to expectant management. The investigators will follow the women with clinical investigations after 2 and 4 weeks. After two weeks the healing will be measured using the REEDA scale and the women will be asked whether they breastfeed or not. The psychological wellbeing will be measured using the EPDS (Edinburgh Postnatal Depression Scale).

After four weeks the above will be done again as well as collecting of the daily pain diary that the women have filled in since being included in the trial.

After one year the women will be seen again and the investigators will do a clinical investigation including ultrasound of the perineal body, measurement of the perineal body, POP-Q ( Pelvic Organ Prolapse Quantification System) as well as multiple validated scales as EPDS, FSFI ( Female Sexual Function Index), PFIQ (Pelvic Floor Impact Questionnaire) and PFDI (Pelvic Floor Distress Inventory). These scales will help the investigators to find out if the women have moderate to much trouble with vaginal wideness and/ or moderate to much problems during defecation and therefore, if the perineal body is palpated smaller than 2 cm, there will be indication for a perineal reconstruction.

The primary outcome will be to investigate whether early resuturing is reducing the need of a later secondary reconstruction of the perineal body compared with conservative management concerning dehisced perineal wounds.

The secondary outcomes will be to investigate whether early resuturing is reducing the risk of having symptoms from the perineum and/or sexual problems one year after delivery.

The healing of the wound and the estimated pain will be compared between the two groups.

Certain questions concerning secondary fear of childbirth will also be asked and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18 years old who had a vaginal delivery and suffered from a perineal rupture, grade 2 (spontaneous or episiotomy).
* No longer than two weeks has passed since delivery.
* The woman must be able to give informed consent.

Exclusion Criteria:

* Perineal rupture grade 3 and 4.
* Woman suffering from connective tissue disease.
* Ongoing treatment with oral cortisone or other immunosuppressive disease.
* Diabetes treated with insulin.
* Suspicion of occult damage of the anal sphincter.
* Earlier surgery of the perineum.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Need of late perineal reconstruction | One year
  Digital palpation of the perineal body and assessment of thickness. POP-Q score; nine points in the vagina are identified. The hymen is the reference point to which the other points are compared. The prolapsed organs are measured in centimeters to the hymen. The measurements are taken when the Valsalva maneuver is performed by the woman.
  Anovaginal distance using perineal ultrasound. Validated scales to identify specific symptoms from the perineum and to identify the feeling of vaginal wideness and the need for digital assistance during defecation.
  PFDI 20- short form-version of pelvic floor distress inventory FSFI - female sexual function index PFIQ - pelvic floor impact questionnaire

SECONDARY OUTCOMES:
Pelvic floor symptoms and the impact on quality of life | One year
  The PFDI 20 is both a symptom inventory and a measure of the degree of bother and distress (quality-of-life) caused by pelvic floor symptoms. It includes 20 questions and 3 scales. The 3 scales include questions taken from the following widely used outcome measures: Urinary Distress Inventory - 6 questions, Pelvic Organ Prolapse Distress Inventory - 6 questions, and Colorectal-Anal Distress Inventory - 8 questions. Each of the 3 scales is scored from 0 (least distress) to 100 (greatest distress). The sum of the scores of these 3 scales serves as the overall summary score of the PFDI-20 and ranges from 0 - 300.
Pelvic floor symptoms and the impact on quality of life | One year
  The PFIQ-7 is used to assess life impact in women with pelvic floor disorders. It consists of 3 scales of 7 questions each taken from the Urinary Impact Questionnaire, the Pelvic Organ Prolapse Impact Questionnaire, and the Colorectal-Anal Impact Questionnaire. The 3 scales are scored from 0 (least impact) to 100 (greatest impact) and an overall summary score (0 to 300).
Sexual function | One year
  The FSFI comprises of a 19 item questionnaire focused on sexual functioning. There are six domains assessed. The subject is advised to consider each of the questions in the context of the last 4 weeks. The answer choices in the FSFI carry a number of points and are summed to obtain six domain scores and an overall score. For the latter here is a threshold at 26.55 which means that all values below are classed as indicating female sexual dysfunction (FSD).
Wound healing | 2 weeks
  REEDA ( Redness, Oedema, Ecchymosis, Discharge, Approximation) scale contains five criteria namely redness, edema, ecchymosis, discharge, and approximation of the wound edges, each receiving a score between 0 and 3. Thus, the total score could range from 0 to 15, with lower scores representing better-wound healing.
Wound healing | 4 weeks
  REEDA scale contains five criteria namely redness, edema, ecchymosis, discharge, and approximation of the wound edges, each receiving a score between 0 and 3. Thus, the total score could range from 0 to 15, with lower scores representing better-wound healing.
Pain intensity measure: NRS | From randomization to 4 weeks after.
  Self reported daily pain intensity. NRS ( numeric rating scale), each day is scored 0-10 ( 0= no pain, 10= pain as bad as can be).
Secondary fear of childbirth | One year.
  One question concerning fear of giving birth in the future will be asked: "What kind of delivery method would you prefer if getting pregnant again in the future, vaginal delivery or planned c-section?". W-DEQ B (Wijma Delivery Expectancy Questionnaire) is a questionnaire measuring the fear of giving birth after delivering. The questionnaire consists of 33 questions, every question has a score from 1-6. The higher score, the higher is the fear of giving birth.
Affected breastfeeding | 2 weeks
  The participant will be asked whether she breastfeeds or not.
Affected breastfeeding | 4 weeks
  The participant will be asked whether she breastfeeds or not.
Psychological wellbeing | 4 weeks
  EPDS- Edinburgh Postnatal Depression Scale . EPDS is a self assessment questionnaire consisting of ten statements and the respondent is asked about her feelings the last seven days. The answers are scored from 0-3 which gives an endpoint from 0-30. In Sweden women are said to have depressive symptoms after delivery if scoring 12 or higher.
Psychological wellbeing | One year.
  EPDS- Edinburgh Postnatal Depression Scale . EPDS is a self assessment questionnaire consisting of ten statements and the respondent is asked about her feelings the last seven days. The answers are scored from 0-3 which gives an endpoint from 0-30. In Sweden women are said to have depressive symptoms after delivery if scoring 12 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Ek, PhD, MD, Principal Investigator — Department of Obstetrics and Gynecology, Stockholm South General Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Stockholm South General Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No